CLINICAL TRIAL: NCT00895115
Title: A Randomized Study to Investigate the Presence of Tocopherol Metabolites in the Prostate
Brief Title: Vitamin E Supplements in Preventing Cancer in Patients at Risk of Prostate Cancer or Who Have Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 120802; P30CA072720 (NIH); CDR0000639070 (Other: NIH)
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm I (Sham Comparator): Patients receive no supplementation.
  Interventions: Procedure: sham intervention
- Arm II (Experimental): Patients receive oral high γ-tocopherol vitamin E supplementation once daily for 1 week.
  Interventions: Dietary Supplement: vitamin E
- Arm III (Experimental): Patients receive oral high γ-tocopherol vitamin E supplementation once daily for 2 weeks.
  Interventions: Dietary Supplement: vitamin E

INTERVENTIONS:
Dietary Supplement: vitamin E — Given once daily
  Arms: Arm II; Arm III
Procedure: sham intervention — No supplementation
  Arms: Arm I

SUMMARY:
RATIONALE: Vitamin E supplements may stop or delay the development of prostate cancer in patients who are at risk of prostate cancer or who have prostate cancer. It is not yet known which vitamin E regimen is more effective in preventing prostate cancer.

PURPOSE: This randomized phase I trial is comparing vitamin E supplement regimens to see how well they work in preventing cancer in patients at risk of prostate cancer or who have prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of tocopherol supplementation on plasma and urine levels of α-, γ-, and δ-tocopherols, PSA, and prostaglandin E_2 by comparing the blood and urine samples collected before and after the supplementation in patients with prostate cancer.
* Test the hypothesis that the supplementation reduced oxidative and nitrosative stress by measuring plasma levels of F_2-isoprostane, C-reactive protein, and 3-nitrotyrosine as well as urinary levels of 8-hydroxy-2-deoxyguanosine (8-OHdG).
* Determine the levels of α-, γ-, and δ-tocopherols in prostate tissues and analyze immunohistochemically (IHC) for cell proliferation, apoptosis, cyclooxygenase-2, 8-OHdG, and 3-nitropyrosine levels in prostate cancer/tissue slides.

OUTLINE: Patients are randomized into 1 of 3 arms.

* Arm I: Patients receive no supplementation.
* Arm II: Patients receive oral high γ-tocopherol vitamin E supplementation once daily for 1 week.
* Arm III: Patients receive oral high γ-tocopherol vitamin E supplementation once daily for 2 weeks.

Blood, urine, and tissue samples are collected periodically and analyzed for oxidative/nitrosative stress and other markers (i.e., F2-isoprostane, 8-OHdG, 3-nitrotyrosine, prostaglandin E2, C-reactive protein, and PSA), biomarkers in prostate tumors and nontumorous tissues (i.e., 8-OHdG, 3-nitrotyrosine, and cyclooxygenase-2) by IHC, and pharmacokinetics by high-performance liquid chromatography.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets one of the following criteria:

  * Abnormal digital rectal examination or abnormal prostate specific antigen (> 4.0 ng/mL)
  * Obstructing prostate
  * Biopsy-proven prostate cancer
* Scheduled to undergo prostate surgery (i.e., transurethral prostatectomy or prostatectomy)

PATIENT CHARACTERISTICS:

* No uncontrolled diabetes, uncontrolled blood pressure, chronic congestive heart failure, or history of renal insufficiency
* No personal or family history of a bleeding disorder
* No known history of problems absorbing dietary fats (e.g., Crohn's disease, cystic fibrosis)

PRIOR CONCURRENT THERAPY:

* More than 2 weeks since prior NSAIDs or corticosteroids
* No concurrent supplementation of vitamin E (a multivitamin containing ≤ 60 IU of vitamin E is allowed)
* No concurrent colestipol or orlistat
* No concurrent warfarin or dicumarol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Effect of tocopherol supplementation on plasma and urine levels of α-, γ-, and δ-tocopherols, PSA, and prostaglandin E2 | 4 years
Oxidative stress and nitrosative stress as assessed by plasma levels of F2-isoprostane, C-reactive protein, and 3-nitrotyrosine as well as urinary levels of 8-hydroxy-2-deoxyguanosine (8-OHdG) | 4 years
Levels of α-, γ-, and δ-tocopherols in prostate tissues and cell proliferation, apoptosis, cyclooxygenase-2, 8-OHdG, and 3-nitropyrosine levels as assessed by IHC | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Susan Goodin, PharmD, FCCP, BCOP, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States